CLINICAL TRIAL: NCT05503550
Title: Pre-Approval Access Single Patient Request Treatment for Talquetamab for Treating Physician Use in Relapsed or Refractory Multiple Myeloma
Brief Title: Pre-Approval Access Single Patient Request for Talquetamab in Relapsed or Refractory Multiple Myeloma
Status: No longer available | Type: Expanded Access
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR109169; 64407564MMY4002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-08-12; First posted 2022-08-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — talquetamab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Talquetamab — Talquetamab will be administered subcutaneously (SC).
  Other Names: JNJ-64407564

SUMMARY:
The purpose of this pre-approval access program is to provide talquetamab for the treatment of participants with relapsed or refractory multiple myeloma.

Min Age: 18 Years
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC